CLINICAL TRIAL: NCT07195981
Title: EFFECT OF IMMERSIVE VIRTUAL REALITY ON PAIN, PROPIOCEPTION AND BALANCE IN CERVICAL RADICULOPATHY PATIENTS
Brief Title: VIRTUAL REALITY IN CERVICAL RADICULOPATHY PATIENTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005940
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received the selected physical therapy program in addition to virtual reality using Oculus glasses.
  Interventions: Device: virtual reality; Other: selected physical therapy
- control group (Experimental): selected physical therapy program only
  Interventions: Other: selected physical therapy

INTERVENTIONS:
Device: virtual reality — The virtual reality (VR) technology is defined as a system that allows users to interact with images and sounds in a virtual environment, which can stimulate responses and provide real-time feedback concerning their performance.
  Arms: study group
Other: selected physical therapy — selected physical therapy program only included: (Therapeutic Ultrasound device, Transcutaneous Electrical Nerve Stimulation (TENS) and Hot packs)

SUMMARY:
PURPOSE: to investigate the effect of immersive virtual reality on pain, proprioception, and balance in cervical radiculopathy patients BACKGROUND: Cervical radiculopathy (CSR) is a disabling condition that significantly impairs a person's ability to function physically, The application of virtual reality (VR) in rehabilitation therapy offers new possibilities. In addition to the neck-specific sensorimotor training, which appears to improve neck mobility.

DETAILED DESCRIPTION:
Fourty two participants with unilateral cervical radiculopathy. from both sexes were participated in this study. The patients were randomly divided into two equal groups; Study group (22 patients): received the selected physical therapy program in addition to virtual reality using Oculus glasses. (22 patients): received receive a selected physical therapy program only (Therapeutic Ultrasound device, Transcutaneous Electrical Nerve Stimulation (TENS) and Hot packs) (12 sessions) three times per week. The evaluation methods by VR ,CROM Device ,Neck disability scale, VAS, joint position error test .

ELIGIBILITY:
Inclusion Criteria:

* Fourty two participants with unilateral cervical radiculopathy.
* Participants are complaining of neck pain radiating unilaterally down to one arm.
* Their ages range from 35-50 years.
* They are referred by a neurologist with a diagnosis of unilateral cervical radiculopathy.

Exclusion Criteria:

* 1) Cervical myelopathy. 2) Patients with previous cervical surgery. 3) Inflammatory diseases such as rheumatoid arthritis or ankylosing spondylitis 4) Any other musculoskeletal disorders of the spine or upper extremity.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Biodex balance system | six week
  The Biodex balance system considered a reliable evaluation tool for balance include overall stability index
Neck Proprioception | six week
  Neck Proprioception by cervical joint position error via Overhead Laser Pointer

SECONDARY OUTCOMES:
Cervical range of motion (CROM) goniometer device measurements | six week
  The CROM is an inclinometers system with a gravitational reference that is suitable for evaluating the active cervical spine movements in different direction
Neck disability index | six week
  The NDI is a validated self-report questionnaire to detect the level at which the neck pain
Visual analogue scale for pain | six week
  The VAS-p is a method for measuring the intensity of pain on a horizontal straight line of fixed length (10 cm)

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 university, Giza, Giza Governorate, Egypt